CLINICAL TRIAL: NCT07350200
Title: XEN Glaucoma Implant for the Management of Operated Uncontrolled Glaucoma: Results and Complications During a Long-Term Follow-Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5/WIM/2021
Record Dates: First submitted 2025-12-15; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2014-12

CONDITIONS: Glaucoma
Keywords: Glaucoma; XEN glaucoma implant; Uncontrolled Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XEN Glaucoma Implant for the Management of Operated Uncontrolled Glaucoma (Experimental): Group of patients, who underwent XEN implantation and had a history of previous unsuccessful antiglaucoma procedures, and who were subject to surgeries performed by the same experienced surgeon.
  Interventions: Procedure: XEN implantation

INTERVENTIONS:
Procedure: XEN implantation — The surgeon used the ab interno or ab externo technique for XEN implantation. In cases where only the lower quadrants were accessible, the ab externo access was the technique of choice. All treatments were performed with 40 micrograms of mitomycin C, which was injected under the conjunctiva at least 6mm from the corneal limbus in the projection of the future filtering bleb. If a clinically significant cataract was also observed in a phakic patient, the patient qualified for a combined procedure with phacoemulsification and implantation of an artificial intraocular lens.

SUMMARY:
XEN Glaucoma Implant for the Management of Operated Uncontrolled Glaucoma: Results and Complications During a Long-Term Follow-Up

DETAILED DESCRIPTION:
Purpose of the study is to analyze the surgical and refractive outcomes of XEN glaucoma implant, a minimally invasive surgical device for the treatment of operated uncontrolled glaucoma. Intraocular pressure change, best corrected visual acuity, change in glaucoma medications, frequency of slit lamp revision procedures, and frequency of secondary glaucoma surgeries were the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* presence of OUG, defined as prior treatment with surgical or cyclodestructive procedures
* failure to achieve target IOP with maximally tolerated topical IOP-lowering treatment or intolerance to drugs
* both primary and secondary open- and closed-angle glaucoma cases
* presence of healthy mobile conjunctiva in at least one quadrant and bestcorrected visual acuity

Exclusion Criteria:

* presence of clinically significant inflammation or infection within 30 days before surgery, history of corneal refractive surgery, corneal deposits or haze preventing intraoperative viewing of the anterior chamber, presence of an anterior chamber lens, advanced age-related macular degeneration (AMD), known or suspected allergy or sensitivity to porcine products or glutaraldehyde, pregnant or nursing women, and lack of consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
IOP | through study completion, an average of 5 years
  Intraocular Pressure
BCVA | through study completion, an average of 5 years
  The change of best- corrected visual acuity
Visual Field | through study completion, an average of 5 years
  Visual Field of the mean defect

SECONDARY OUTCOMES:
Medications | through study completion, an average of 5 years
  Median number of patients who took medications before surgery and up until the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Military Institute of Medicine - National Research Institute, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No